CLINICAL TRIAL: NCT07202715
Title: Efficacy of CBT Based C.A.T Project for Pakistani Adolescents With Anxiety Disorders- A Pilot Randomized Control Trial.
Brief Title: RCT of CBT Based C.A.T Project for Pakistani Adolescents With Anxiety Disorders.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Science and Technology (Other)
Responsible Party: Principal Investigator, Annum Tanweer, Principal Investigator, PhD Scholar, National University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0839
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorder of Adolescence
Keywords: Adolescent Anxiety Disorders, CBT, RCT
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Intervention Model Description: 50 students, who screened postive for anxiety disorders using SCARED screening tool were randomly selected from three randomly selected schools (selected from online PEPRIS List of schools in Rawalpindi) for the study. 50 students were then randomly assigned to either an experimental or waitlist/TAU group.
  16 week CBT based C.A.T Project treatment will be given to the participants in experimental group.
Who Masked: Outcomes Assessor
Masking Description: The outcome measure assesments before, during and after intervention will be completed and assessed by an independent team of 2 clinical psychologists. 3 month Followup assessment will be carried out by independent team of 2 psychologists .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - C.A.T Project Intervention (Experimental): In this group 25 participants will receive C.A.T Project (CBT based treatment for anxious adolecents) intervention program. This is an evidence based 16 week program designed to alleviate the symptoms of anxiety disorder among teenagers. The intervention will be delivered over 16 weeks, with weekly structured and videoptapped sessions involving adolescents and their parents. 14 sessions are delivered to adolescents and 2 sessions are parental sessions. The sessions will be delivered in groups of 3-5 students. The program includes psychoeducation, learing coping skills, enhancing emotional regulation, problem solving, relaxation and exposure exercises. Parents and teachers will be actively engaged througout the program.
  Interventions: Behavioral: CBT Based C.A.T Project- Intervention for Anxious Adolescents.
- Waitlist/TAU Group- no Intervention (No Intervention): 25 participants in the waitlist/TAU group will receive no active intervention during the study period but continued to access routine care/ teacher's guidance as available. After the trial and 3 month followup will end, they will be offered the experimental intervention.
  The waitlist/TAU group will serve as a control condition, allowing researchers to compare the effects of the intervention against participants receiving only standard and usual care.

INTERVENTIONS:
Behavioral: CBT Based C.A.T Project- Intervention for Anxious Adolescents. — The C.A.T Project is a structured, evidence-based intervention grounded in Cognitive Behavioral Therapy (CBT) principles, designed specifically for adolescents experiencing anxiety and related concerns. The core components includes: Psychoeducation, Cognitive Restructuring, Exposure Exercises, Coping Skills Training and Relapse Prevention. This age appropriate intervention will be delivered in Urdu language with culturally appropriate context.
  Arms: Experimental Group - C.A.T Project Intervention

SUMMARY:
Anxiety Disorders are the most prevalent mental health conditions among adolescents. The current randomized control trial aims to assess the efficacy of the C.A.T Project protocol among adolescents aged 14 to 17 years diagnosed with severe to moderate anxiety disorders in school settings. The research explores the impact of the intervention on reducing acute and chronic symptoms of anxiety, academic performance, self concept, overall wellbeing, internalizing and externalizing behaviors among school going adolescents with anxiety concerns. The intervention integrates various components of Cognitive Behavioral Therapy using cognitive restructuring, parental psychoeducation, behavioral activation, problem solving and relaxation exercise. The study had already completed translation and adaptation of the C.A.T Workbook for adolescents in Urdu language and context using Brislin (1976) and WHO (2023) guidelines.

The CBT model is a multifaceted, evidence-based treatment for adolescents diagnosed with various kinds of anxiety disorders. It aims to identify and change unhelpful thought patterns to more helpful thinking leading to positive emotions and behaviors. It also is evidenced to be effective with various levels of severity and comorbidity. In this study, the 16-week intervention will be tested through a randomized waitlist/TAU trial, where 50 participants are be divided into intervention and control arms. In addition to various outcomes, the research also aims to evaluate fidelity, feasibility and acceptability of the protocol at school setting in Pakistan. Post and 3 month follow up will be explored to determine immediate and long-term treatment efficacy.

DETAILED DESCRIPTION:
The current research is a randomized control trial to evaluate the efficacy of the CBT based C.A.T Project for adolescents aged 14-17 years with anxiety disorders. Globally and locally anxiety disorders are one of the most prevalent mental health concerns among adolescents and young adults (WHO, 2025), however in developing concerns it remains underdiagnosed and untreated especially among school going adolescents. The study aims to address this gap by adapting evidence-based resources and implementing them in Pakistani context. In the first phase of the study the C.A.T Workbook (Kendall 1994, 1997) for adolescents was linguistically translated and culturally adapted using WHO (2023) and Brislin (1976) guidelines using procedures like expert panel review, cognitive interviewing and content validity assessment (CVI =0.96).

Integrating Cognitive Behavioral approach, the C.A.T Project for adolescents include the following components: Therapist manual and teen workbook (translated and culturally adapted in Urdu), parental and adolescent psychoeducation, changing adolescent's negative perceptions and cognitions, weekly homework exercises, exposure tasks.

To select participants in the current trial, 3 schools in Rawalpindi, Pakistan were randomly selected from the online PEPRIS List. Adhering to all the ethical requirements of assent and consent from various stakeholders, students were screened for anxiety disorders using standardized and adapted tools. 50 students, who screened postive for anxiety disorders using SCARED screening tool were randomly selected from those selected school for the study. 50 students were then randomly assigned to either an experimental or waitlist/TAU group. Further assessment on outcome measures and standardized diagnostic interviewing using Kiddie SADS protocol was carried out using culturally adapted measures. The intervention is delivered to groups of 3-5 students per session. The intervention is 16 weeklong, with one session per week. 14 sessions are for adolescents while 2 sessions are for their parents. Outcome measures are assessed before, during and post intervention with a 3-month follow-up assessment. These assessments from adolescents, parents and teachers are carried out by an independent team of clinical psychologists to reduce bias. Outcome measures include evaluating acute and chronic symptoms of anxiety in various time points, academic performance, their self-concept, overall mental wellbeing, screentime addiction, physical activity, internalizing and externalizing behaviors like emotional symptom, conduct problems, hyperactivity-inattention, peer problems and prosocial behavior among school going adolescents with anxiety concerns. Overall mental wellbeing of parents and teachers are also noted.

The current study adheres to the CONSORT guidelines for feasibility studies. Keeping in view of the confidentiality and privacy of the participants, each session is video recorded and is evaluated by an independent team of clinical psychologists using standardized feasibility and protocol adherence questionnaires. The result of this study is expected to show the reduction of symptoms of anxiety disorders, improve adolescent's overall mental wellbeing and inform evidence on scalability, practicality and effectiveness of CBT based standard mental health services in school settings.

The description of the study is clear and adheres to the requirements and guidelines of ClinicalTrials.gov. It mentions the purpose, design, methodology and expected findings of the study.

Objectives:

The main objectives of the study are

1. To determine the fidelity, feasibility and acceptability of the CBT based C.A.T Project for adolescents in Pakistani context.
2. To linguistically translate and culturally adapt the CBT based C.A.T Project Workbook for Project for use with Urdu-speaking adolescents in Pakistan.
3. To evaluate the efficacy of C.A. T Project treatment compared to standard care alleviate symptoms of anxiety disorders among adolescents in school setting.
4. To assess the impact of C.A. T Project intervention on academic performance, internalizing and externalizing behaviors, overall wellbeing and self-concept among adolescents diagnosed with anxiety disorders.
5. To investigate the impact of C.A.T Project intervention on screentime addiction of adolescents diagnosed with anxiety disorders.
6. To evaluate the maintenance of treatment effects in adolescents diagnosed with anxiety disorders through 3-month post treatment follow up.

Hypothesis:

1. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in their acute and chronic symptoms of anxiety disorders from their baseline and as compared to the waitlist/TAU group.
2. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in internalizing and externalizing behaviors, as compared to the waitlist/TAU group.
3. Parents and adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in overall mental wellbeing as compared to the waitlist/TAU group.
4. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant reduction in experiencing screentime addiction as compared to thewaitlist/TAU group.
5. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in physical activity as compared to the waitlist/TAU group.
6. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in their self-concept as compared to the waitlist/TAU group.
7. Teachers and Parental overall mental wellbeing will have a statistically significant relationship with overall mental wellbeing of the Adolescents with Anxiety Disorder.
8. Adolescents with Anxiety Disorder who receive CBT based C.A.T Project intervention will demonstrate statistically significant improvement in their acute and chronic symptoms of anxiety disorders and outcome measures from their baseline and as compared to the waitlist/TAU group after 3 month followup.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 14-17-year-old in school setting, who score above the cutoff score (25) on SCARED (Screening for Child Anxiety Related Disorders) for Child and/or Parent version become part of this study. Further diagnostic interviewing is carried out to explore severity and comorbidity using structured and urdu translated Kiddie SADS-PL diagnotic interviewing protocol.

Exclusion Criteria:

* Students who score below the cutoff score of 25 on SCARED (Screening for Child Anxiety Related Disorders) assessment for Child and/or Parent version are not part of the study. Students who were screened for Neurodevelopmental concerns like ADHD and ASD using Kiddie SADS- PL interview protocols are not considered to be part of the study. In addition, participants who are currently undergoing medical/psychological treatment for their anxiety related concerns are not part of this study.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders | Pretesting phase, 4 month and 3 month followup
  The Screen for Child Anxiety Related Emotional Disorders (SCARED) scale will be used with adolescents. The scale ranges from 0 to 82, with higher scores indicating greater severity of anxiety symptoms (i.e., a worse outcome)
Fear Survey Schedule for Children-Revised | Pretesting phase, 4 months and 3 month followup
  The Fear Survey Schedule for Children-Revised (FSSC-R), Urdu version will be used with adolescents. The scale ranges from 80 to 240, with higher scores indicating greater severity of fears (i.e., a worse outcome).
Diagnostic Assesment on Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime | Pretesting phase, 4 month and 3 month followup
  The Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version (K-SADS-PL), Urdu version, will be used with adolescents. This is a semi-structured diagnostic interview rather than a numerical scale, so it does not have a minimum or maximum score. Outcomes are reported as the presence or absence of psychiatric diagnoses based on DSM criteria, with endorsement of a diagnosis reflecting a worse outcome.
Childhood Anxiety Sensitivity Index | Pretesting phase, 4 month and 3 month followup
  The Childhood Anxiety Sensitivity Index (CASI) will be used with adolescents. The scale ranges from 18 to 54, with higher scores indicating greater anxiety sensitivity (i.e., a worse outcome).

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Pretesting, 4 months and 3 month followup
  The Strengths and Difficulties Questionnaire (SDQ) has five subscales: Emotional, Conduct, Hyperactivity, Peer, and Prosocial (all 0-10). Higher scores on Emotional, Conduct, Hyperactivity, and Peer indicate more problems (worse outcome), while higher Prosocial scores indicate better outcomes. Composite scores include Total Difficulties (0-40), Internalizing (0-20), and Externalizing (0-20), where higher scores reflect worse outcomes.
Adolescent's Self-Concept Short Scale | Pretesting, 4 months and 3 month followup
  e measure consists of 30 items with a total score range from 30 to 150, where higher scores reflect a more positive self-concept and lower scores indicate a poorer self-concept. Factor analysis of the Urdu version identified four subscales: Anxiety (8 items; range 8-40), where higher scores indicate greater anxiety and thus a less adaptive self-concept; Physical Appearance (8 items; range 8-40), where higher scores reflect a more positive perception of appearance; Behavior (6 items; range 6-30), where higher scores indicate more positive self-perceived behavior; and Intellectual Status (4 items; range 4-20), where higher scores reflect stronger perceived intellectual abilities. Together, these domains provide both a total score and domain-specific insights into adolescents' self-concept.
WHO-5 Well-Being Index for Adolescents | Pretesting, 4 months and 3 month followup
  The World Health Organization-Five Well-Being Index (WHO-5) will be used with adolescents. This self-report measure consists of 5 positively worded items rated on a 6-point Likert scale (0 = "at no time" to 5 = "all of the time"), giving a raw score range of 0 to 25. The raw score is commonly multiplied by 4 to yield a standardized score ranging from 0 to 100. Higher scores indicate better subjective well-being, while lower scores reflect poorer well-being and may be indicative of risk for depression.
Smartphone Addiction Scale - Short Version | 4 months and 3 month followup
  his measure consists of 10 items, each rated on a 6-point Likert scale from 1 ("strongly disagree") to 6 ("strongly agree"), yielding a total score range of 10 to 60. Higher scores indicate greater severity of smartphone addiction (worse outcome), while lower scores reflect healthier smartphone use.
Competence and Adherence Scale for CBT (CAS-CBT) | 4 months
  A standardized tool evaluating therapist competence and treatment adherence in delivering CBT for youth anxiety.
Summary Therapist Feedback | 4 months
  Structured forms for therapists to provide consolidated feedback on session progress and client engagement.
Manual Rating Form | 4 months
  checklist-based tool assessing fidelity and adherence to treatment manuals during therapy sessions.
Rates of Perceived Benefits from Treatment | 4 months
  Self reported ratings of the extent to which therapy outcomes are seen as helpful or beneficial.
Weekly Therapist Feedback Form | 4 month
  Ongoing therapist-completed form capturing weekly observations of client progress, engagement, and challenges.
Physical Activity (Demographic Variable) | Pretesting, 4 month and 3 month followup
  Participants will be asked to self-report the average number of hours per week they engage in physical activity (e.g., sports, exercise, walking). Responses will be recorded as a continuous variable in hours, providing an estimate of overall activity level. engaging in at least 60 minutes per day (≥7 hours per week) of moderate-to-vigorous physical activity is considered meeting the recommended guideline, while reporting less than this threshold will be classified as insufficient physical activity.
Academic performance (Demographic Variable) | Pretesting, 4 month and 3 month followup
  Participants will be asked to self-report their most recent academic performance (e.g., percentage marks, grade point average, or grade equivalent). Responses will be recorded as a continuous variable (percentage or GPA) where available. For interpretation, scores may also be categorized according to conventional academic performance bands (e.g., High: ≥80%, Moderate: 60-79%, Low: <60%) to facilitate comparison across participants.
WHO-5 Well-Being Index for parent | Pretesting phase, 4 month and 3 month followup
  The World Health Organization-Five Well-Being Index (WHO-5) will be used with adolescents. This self-report measure consists of 5 positively worded items rated on a 6-point Likert scale (0 = "at no time" to 5 = "all of the time"), giving a raw score range of 0 to 25. The raw score is commonly multiplied by 4 to yield a standardized score ranging from 0 to 100. Higher scores indicate better subjective well-being, while lower scores reflect poorer well-being and may be indicative of risk for depression in their parent
WHO-5 Well-Being Index for teacher | Pretesting phase, 4 month and 3 month followup
  The World Health Organization-Five Well-Being Index (WHO-5) will be used with adolescents. This self-report measure consists of 5 positively worded items rated on a 6-point Likert scale (0 = "at no time" to 5 = "all of the time"), giving a raw score range of 0 to 25. The raw score is commonly multiplied by 4 to yield a standardized score ranging from 0 to 100. Higher scores indicate better subjective well-being, while lower scores reflect poorer well-being and may be indicative of risk for depression in their teacher.

CONTACTS AND LOCATIONS:
Overall Officials: Annum Tanweer, Principal Investigator — School of Social Sciences and Humanities, NUST, Islamabad
Locations (3):
- Pakistan (3):
  - CRM School system, Rawalpindi, Punjab Province
  - Amblem School System, Rawalpindi, Punjab Province
  - Spangle House School, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Keeping in view of the confidentiality